CLINICAL TRIAL: NCT04837157
Title: Evaluation of the Safety of ATLAS 2030 in the Application of Robot-assisted Physical Therapy to Children With Neuromuscular Diseases Phase I
Brief Title: Evaluation of the Exoskeleton ATLAS 2030 as Robot-assisted Physical Therapy to Children With Neuromuscular Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MarsiBionics (Industry)
Collaborators: Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ATLAS2030ENM-I
Record Dates: First submitted 2020-11-03; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Cerebral Palsy; SMA II; Neuromuscular Diseases
Keywords: Exoskeleton; robot-assisted; physical therapy; ATLAS
MeSH Terms: conditions — Cerebral Palsy; Spinal Muscular Atrophies of Childhood; Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): 9 treatment sessions will be performed with the ATLAS2030 exoskeleton. The rehabilitation sessions last approximately 90 minutes. Two sessions are scheduled per week, for two weeks.
  Interventions: Device: Exoskeleton rehabilitation

INTERVENTIONS:
Device: Exoskeleton rehabilitation — The participants will perform physical therapy with the ATLSA2030 device, for 90 minutes per session.
  Other Names: ATLAS2030; ATLAS; robot-assisted therapy

SUMMARY:
This study aims to evaluate the safety, usability and acceptability of a motorized mobility assistance exoskeleton. The protocol explores the use of the motorized device during static and dynamic rehabilitation sessions focused on walking and functional activities, with the expectation of evaluating the safety and usability of the device in the population studied. The protocol has been focused on defining how the device can be used appropriately in this population in a safe and effective manner by rehabilitation specialists. The study also aims to assess the safety of clinical staff who implement the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Maximum user weight of 35 kg
* Thigh length (distance from the greater trochanter to the lateral condyle of the tibia) from 24 cm to 40 cm.
* Leg length (distance from the lateral condyle of the tibia to the lateral malleolus) from 23 to 39 cm.
* Pelvis width (between greater trochanters) from 24 to 35 cm.
* Ability to achieve ankle dorsiflexion to 90˚
* 20º or more hip flessum.
* 20º or more knee flessum.
* No allergies to any of the ATLAS materials: cotton, nylon, polyester, polyamide, polyethylene or propylene.
* Informed consent signed by legal guardians.
* Confirmed diagnosis of cerebral palsy or neuromuscular disease affecting walking ability at early development stages
* Stable medical condition with no changes in disease-specific medication in the last 6 months, and additional medication in the last month.
* Patient being followed according to the recommended standards for his or her illness
* Ability to maintain, spontaneously or with a brace, the head and trunk while standing and walking.
* No need for daytime ventilation (have an oxygen saturation and PCO2 with normal ambient oxygen
* Score on the FAC scale between 1 and 4 points
* Not being able to walk without assistance

Exclusion Criteria:

* Patient's inability to follow simple instructions and/or communicate discomfort.
* Invasive or non-invasive daytime ventilation.
* Orthostatic hypotension.
* 20º or more hip flessum.
* 20º or more knee flessum
* Scoliosis with a Cobb angle of more than 25º that cannot wear a corset during the test.
* Severe skin injury to the lower extremities.
* Scheduled surgery (spine, extremities) during the period of the study or surgery performed (spine, extremities) in the last 6 months.
* History of fracture without trauma.
* History of traumatic bone fracture in lower limbs or pelvic girdle in the last 3 months
* Not receiving regular standing rehabilitation sessions.
* Absence of control of the head or trunk in an upright position without the possibility of wearing a corset during the use of the exoskeleton
* Refusal of the patient or legal guardian to include the child in the study.
* Skin problems (diseases, allergies, sensitivity ...) that prevent the use of exoskeleton accessories on the skin of patients.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Safety as number of serious device adverse events | after each use of exoskeleton, for 5 weeks
  Presence of a serious device adverse events where the participant or therapist is involved

SECONDARY OUTCOMES:
Safety as presence of adverse events or adverse device events | after each use of exoskeleton, for 5 weeks
  Presence of a device adverse events where the participant or therapist is involved.
Exercises [measured as time per exercise in seconds] | after each use of exoskeleton, for 5 weeks
  Measured as time per event for at each therapy session.
Transfers [measured as time to carry out the transfers in seconds] | At each use of exoskeleton, for 5 weeks
  Measured as time to carry out the transfers
Acceptability [number of participants which discontinue the participation during the trial in relation with the included participants] | At the end of the study, at the 5th week
  Measured as abandon ratio
Accessibility [number of potential participants in relation with the included participants] | At the end of the study, at the 5th week
  Measured as relation between number of participants and number of potential participants which weren't recruited
Fall Prevalence [number of falls during the using of the device] | During the use of the device, for 5 weeks
  Number of falling events ocurred from the participant or therapist
Skin integrity [number of skin injuries related to the device] | before and after each use of exoskeleton, for 5 weeks
  skin integrity measured as the number of skin injuries
Pain [Wong-Baker FACES Pain Rating Scale] | Before and after the use of the device, during 5 weeks
  Pain registered before and after the use of the device, by the participant and therapist. The options are from 1 to 6. A higher score means a worse outcome.
Fatigue [Borg Rating Scale of Perceived Exertion] | Before and after the use of the device, during 5 weeks
  Fatigue registered before and after the use of the device, by the participant and therapist. Measured from 0 to 10, being 0 as fully rested and 10 very tired. A higher score means a worse outcome.
Spasticity [Modified Ashworth Scale] | Before and after the use of the device, during 5 weeks
  Spasticity registered before and after the use of the device
Heart rate [sphygmomanometer] | Before and after the use of the device, during 5 weeks
  Number of heart bets per minute
Physical evaluation [number of physical injuries detected] | Before and after the use of the device, during 5 weeks
  Physical Evaluation as presence of tissue damage
Muscle Strength [measured with Hand Held Dynamometer in N] | At the first day, 3rd week and 5th week
  Muscle Strength measured at hip, knee and ankle muscles
ROM [measured with goniometer] | At the first day, 3rd week and 5th week
  Range of Movement
Functional Mobility [Functional Ambulation Category scale] | At the first day, 3rd week and 5th week
  Functional Mobility with and without the device
System Usability [System Usability Scale] | At the end of the study, 5th week
  Measurement of System's Usability measured by the therapist
User perception of the device [QUEST 2.0 and QUEST 2.1] | At the end of the study, 5th week
  QUEST 2.0 will be assessed by the therapist, and QUEST 2.1 will be assessed by the participant
Distance covered walking [6MWT] | At the first day, 3rd week and 5th week
  6MWT recorded using the device
Device malfunction [as number and type of device malfunction] | During the use of the device, for 5 weeks
  Any device malfunction will be recorded
Particpant's stability [Functional Reach Test] | At the first day, 3rd week and 5th week
  Functional Reach Test
Systolic/Diastolic Pressure [sphygmomanometer] | Before and after the use of the device, during 5 weeks
  Systolic Pressure and Diastolic Pressure measured with sphygmomanometer (measured in mmHg)
Breath Rate [number of breaths per minute] | Before and after the use of the device, during 5 weeks
  Number of breaths per minute
SpO2 [pulse oximeter] | Before and after the use of the device, during 5 weeks
  SpO2 measured as %

CONTACTS AND LOCATIONS:
Locations (1):
- MarsiCare, Arganda, Madrid, Spain

REFERENCES:
- [Derived] Cumplido-Trasmonte C, Ramos-Rojas J, Delgado-Castillejo E, Garces-Castellote E, Puyuelo-Quintana G, Destarac-Eguizabal MA, Barquin-Santos E, Plaza-Flores A, Hernandez-Melero M, Gutierrez-Ayala A, Martinez-Moreno M, Garcia-Armada E. Effects of ATLAS 2030 gait exoskeleton on strength and range of motion in children with spinal muscular atrophy II: a case series. J Neuroeng Rehabil. 2022 Jul 19;19(1):75. doi: 10.1186/s12984-022-01055-x. PMID 35854321